CLINICAL TRIAL: NCT05882578
Title: Effects of Exercise Oncology Intervention in Fitness Capacity and Body Composition in Breast Cancer Survivals
Acronym: WIM_22
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tigers Running Club (Other)
Responsible Party: Principal Investigator, Soraya Casla Barrio, Director of Oncologic Physical Exercise Area and PhD in Exercise Psychology, Tigers Running Club
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WIM_SURVIVALS_22
Record Dates: First submitted 2023-05-22; First posted 2023-05-31 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Cancer Survivors
Keywords: Breast Cancer; Exercise Oncology; Cancer Survivors; Fitness Capacity; Quality of life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: control trial
Masking Description: Doesn´t exist. Patients were allocated depending their preferences
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients will be assessed and screened prior the intervention. After the physical assestment they will attend 2 days a week for the supervised, and controlled sessions of physical exercise, performed in the nature (Retiro park in Madrid). To meassure the intensity of the program, they will use the 1-10 Borg ratio of perceived exertion (RPE).
  Interventions: Other: Oncological physical exercise intervention
- Control Group (Active Comparator): Patients will be asked to mantain an active lifestyle, performing physical activity regularly.
  Interventions: Other: Active Physical Activities intervention

INTERVENTIONS:
Other: Oncological physical exercise intervention — An initial physical assestment where clinical history, body composition, functionality, cardiovascular fitness and quality of life will be tested.
  Patients will be screened and then divided in diferent groups, depending on both their cardiovascular and physical capacity.
  Then they will perform 2 sessions of combined strength and endurance training per week for 16 weeks.
  At the end of the training program, the patients will be assesed to evaluate the changes in their cardiovascular fitness, functionality, body composition and quality of life.
  Arms: Intervention Group
Other: Active Physical Activities intervention — An initial physical assestment where clinical history, body composition, functionality, cardiovascular fitness and quality of life will be tested Patients will be suggested to mantain active physical activities in their daily life.
  At the end of the training program, the patients will be assesed to evaluate the changes in their cardiovascular fitness, functionality, body composition and quality of life.
  Arms: Control Group

SUMMARY:
The goal of this interventional study is to analyze the impact of a supervised oncological exercise intervention in surviving breast cancer patients. The main questions it aims to answer are:

* Evaluate the efectivity of a supervised individualized and adapted oncological physical exercise program in the cardiovascular fitness of the participants.
* Analyze the impact of this intervention in the body composition, functionality and quality of life of the parcitipants

Participants will perform a controlled and adapted program, supervised by an especialized professional during 16 weeks.

Researchers will compare this intervention group, where the supervised program will take place, with a control group, where the patients will perform regular physical activity (non-supervised) to see the changes in the efectivity and impact in cardiovascular fitness, body composition and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with primary, type I to III A/B cancer, with hormonal positive (ER+ and PG+), triple positive (ER+, PG+ y HER2+) or triple negative subtype.
* Women with chemotherapy and radiotherapy phase complete.
* Women with post-surgery phase complete.
* Women that are within 5 years from diagnostic.
* ECOG Score above or equal to 0 or 1.

Exclusion Criteria:

* Submit medical contraindications to physical exercise by their reference doctor.
* Women in state IV o methastasis.
* Pregnant women.
* Meet any of the criteria of the American Thoracic Society (ATS) to perfrom a cardiovascular fitness test.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-04-09 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Cardiovascular fitness | 16 weeks
  Evaluate the effectiveness of the program in the improvement of the cardiovascular capacity in breast cancer survivors (looking for a difference of 3,49 ml/kg/min of oxigen consumption), using a submaximal cardiovascular test.

SECONDARY OUTCOMES:
Body composition | 16 weeks
  Analyze the effect of the oncologic physical exercise program in the body weight, the body mass index (BMI), percentages in body fat, abdominal fat, fat free mass, bone mass and total body water in breast cancer survivors.
Physical functionality | 16 weeks
  Know the impact of the oncologic physical exercise program in the physical functionality of the patients.
Exercise adherence | 16 weeks
  Measure the level of adherence to the oncologic physical exercise program, registering the assistance to the sessions.
Physical activity Levels | 16 weeks
  Evaluate the effect of the intervention in the physical activity levels performed by the patients.
Fatigue levels | 16weeks
  Evaluate the impact of the physical exercise program in the fatigue levels of the participants.
Quality of life and health | 16 weeks
  Evaluate the impact of the oncological physical exercise program in the quality of life of the patients in relation with their health.
Anxiety and depression levels | 16 weeks
  Analyze the impact of the oncologic physical exercise program in the anxiety and depression levels of the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Soraya Casla-Barrio, PhD, Principal Investigator — Tigers Running Club; Helios Pareja-Galeano, PhD, Study Chair — Universidad Autonoma de Madrid; Mónica Castellanos, MSc, Study Chair — Tigers Running Club; Jaime Pérez-Vélez, BSc, Study Chair — Tigers Running Club
Locations (1):
- Tigers Running Club, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
The information will be shared with the patients after the completion of every test.
  This information will be shared only with the participant researchers of this study.

REFERENCES:
- [Background] Runowicz CD, Leach CR, Henry NL, Henry KS, Mackey HT, Cowens-Alvarado RL, Cannady RS, Pratt-Chapman ML, Edge SB, Jacobs LA, Hurria A, Marks LB, LaMonte SJ, Warner E, Lyman GH, Ganz PA. American Cancer Society/American Society of Clinical Oncology Breast Cancer Survivorship Care Guideline. CA Cancer J Clin. 2016 Jan-Feb;66(1):43-73. doi: 10.3322/caac.21319. Epub 2015 Dec 7. PMID 26641959
- [Background] Wang H, Mao X. Evaluation of the Efficacy of Neoadjuvant Chemotherapy for Breast Cancer. Drug Des Devel Ther. 2020 Jun 18;14:2423-2433. doi: 10.2147/DDDT.S253961. eCollection 2020. PMID 32606609
- [Background] Fisusi FA, Akala EO. Drug Combinations in Breast Cancer Therapy. Pharm Nanotechnol. 2019;7(1):3-23. doi: 10.2174/2211738507666190122111224. PMID 30666921
- [Background] Nicolazzi MA, Carnicelli A, Fuorlo M, Scaldaferri A, Masetti R, Landolfi R, Favuzzi AMR. Anthracycline and trastuzumab-induced cardiotoxicity in breast cancer. Eur Rev Med Pharmacol Sci. 2018 Apr;22(7):2175-2185. doi: 10.26355/eurrev_201804_14752. PMID 29687878
- [Background] Minotti G, Menna P, Salvatorelli E, Cairo G, Gianni L. Anthracyclines: molecular advances and pharmacologic developments in antitumor activity and cardiotoxicity. Pharmacol Rev. 2004 Jun;56(2):185-229. doi: 10.1124/pr.56.2.6. PMID 15169927
- [Background] Kotamraju S, Chitambar CR, Kalivendi SV, Joseph J, Kalyanaraman B. Transferrin receptor-dependent iron uptake is responsible for doxorubicin-mediated apoptosis in endothelial cells: role of oxidant-induced iron signaling in apoptosis. J Biol Chem. 2002 May 10;277(19):17179-87. doi: 10.1074/jbc.M111604200. Epub 2002 Feb 20. PMID 11856741
- [Background] Bikiewicz A, Banach M, von Haehling S, Maciejewski M, Bielecka-Dabrowa A. Adjuvant breast cancer treatments cardiotoxicity and modern methods of detection and prevention of cardiac complications. ESC Heart Fail. 2021 Aug;8(4):2397-2418. doi: 10.1002/ehf2.13365. Epub 2021 May 5. PMID 33955207
- [Background] Padegimas A, Clasen S, Ky B. Cardioprotective strategies to prevent breast cancer therapy-induced cardiotoxicity. Trends Cardiovasc Med. 2020 Jan;30(1):22-28. doi: 10.1016/j.tcm.2019.01.006. Epub 2019 Jan 29. PMID 30745071
- [Background] Cardinale D, Iacopo F, Cipolla CM. Cardiotoxicity of Anthracyclines. Front Cardiovasc Med. 2020 Mar 18;7:26. doi: 10.3389/fcvm.2020.00026. eCollection 2020. PMID 32258060
- [Background] Armenian SH, Xu L, Ky B, Sun C, Farol LT, Pal SK, Douglas PS, Bhatia S, Chao C. Cardiovascular Disease Among Survivors of Adult-Onset Cancer: A Community-Based Retrospective Cohort Study. J Clin Oncol. 2016 Apr 1;34(10):1122-30. doi: 10.1200/JCO.2015.64.0409. Epub 2016 Feb 1. PMID 26834065
- [Background] Abdel-Qadir H, Austin PC, Lee DS, Amir E, Tu JV, Thavendiranathan P, Fung K, Anderson GM. A Population-Based Study of Cardiovascular Mortality Following Early-Stage Breast Cancer. JAMA Cardiol. 2017 Jan 1;2(1):88-93. doi: 10.1001/jamacardio.2016.3841. PMID 27732702
- [Background] Cardinale D, Colombo A, Bacchiani G, Tedeschi I, Meroni CA, Veglia F, Civelli M, Lamantia G, Colombo N, Curigliano G, Fiorentini C, Cipolla CM. Early detection of anthracycline cardiotoxicity and improvement with heart failure therapy. Circulation. 2015 Jun 2;131(22):1981-8. doi: 10.1161/CIRCULATIONAHA.114.013777. Epub 2015 May 6. PMID 25948538
- [Background] Jones LW, Eves ND, Haykowsky M, Freedland SJ, Mackey JR. Exercise intolerance in cancer and the role of exercise therapy to reverse dysfunction. Lancet Oncol. 2009 Jun;10(6):598-605. doi: 10.1016/S1470-2045(09)70031-2. PMID 19482248
- [Background] Hurria A, Jones L, Muss HB. Cancer Treatment as an Accelerated Aging Process: Assessment, Biomarkers, and Interventions. Am Soc Clin Oncol Educ Book. 2016;35:e516-22. doi: 10.1200/EDBK_156160. PMID 27249761
- [Background] Jones LW, Courneya KS, Mackey JR, Muss HB, Pituskin EN, Scott JM, Hornsby WE, Coan AD, Herndon JE 2nd, Douglas PS, Haykowsky M. Cardiopulmonary function and age-related decline across the breast cancer survivorship continuum. J Clin Oncol. 2012 Jul 10;30(20):2530-7. doi: 10.1200/JCO.2011.39.9014. Epub 2012 May 21. PMID 22614980
- [Background] Adams MJ, Lipsitz SR, Colan SD, Tarbell NJ, Treves ST, Diller L, Greenbaum N, Mauch P, Lipshultz SE. Cardiovascular status in long-term survivors of Hodgkin's disease treated with chest radiotherapy. J Clin Oncol. 2004 Aug 1;22(15):3139-48. doi: 10.1200/JCO.2004.09.109. PMID 15284266
- [Background] Foulkes SJ, Howden EJ, Bigaran A, Janssens K, Antill Y, Loi S, Claus P, Haykowsky MJ, Daly RM, Fraser SF, LA Gerche A. Persistent Impairment in Cardiopulmonary Fitness after Breast Cancer Chemotherapy. Med Sci Sports Exerc. 2019 Aug;51(8):1573-1581. doi: 10.1249/MSS.0000000000001970. PMID 30829962
- [Background] Brubaker P, Jensen A, Jordan J, Lamar Z, Mihalko S, Haykowsky M, Jones L, D Agostino R Jr, Kitzman D, Reding K, Hundley WG. Exercise Capacity Is Reduced in Cancer Survivors Previously Treated With Anthracycline-Based Chemotherapy Despite a Preserved Cardiac Output Response. JACC Cardiovasc Imaging. 2019 Nov;12(11 Pt 1):2267-2269. doi: 10.1016/j.jcmg.2019.05.016. Epub 2019 Jul 17. No abstract available. PMID 31326490
- [Background] Groarke JD, Payne DL, Claggett B, Mehra MR, Gong J, Caron J, Mahmood SS, Hainer J, Neilan TG, Partridge AH, Di Carli M, Jones LW, Nohria A. Association of post-diagnosis cardiorespiratory fitness with cause-specific mortality in cancer. Eur Heart J Qual Care Clin Outcomes. 2020 Oct 1;6(4):315-322. doi: 10.1093/ehjqcco/qcaa015. PMID 32167560
- [Background] Bortolozo HI, Derchain S, Vechin FC, Maginador GF, Santos IS, Torresan R, de Nazare Silva Dos Santos P, Sarian LO, Conceicao MS. Aerobic Fitness is a Predictor of Body Composition in Women With Breast Cancer at Diagnosis. Clin Breast Cancer. 2021 Jun;21(3):e245-e251. doi: 10.1016/j.clbc.2020.10.001. Epub 2020 Oct 9. PMID 34159902
- [Background] Kirkham AA, Bland KA, Sayyari S, Campbell KL, Davis MK. Clinically Relevant Physical Benefits of Exercise Interventions in Breast Cancer Survivors. Curr Oncol Rep. 2016 Feb;18(2):12. doi: 10.1007/s11912-015-0496-3. PMID 26769117
- [Background] Schmidt T, van Mackelenbergh M, Wesch D, Mundhenke C. Physical activity influences the immune system of breast cancer patients. J Cancer Res Ther. 2017 Jul-Sep;13(3):392-398. doi: 10.4103/0973-1482.150356. PMID 28862198
- [Background] Leclerc AF, Foidart-Dessalle M, Tomasella M, Coucke P, Devos M, Bruyere O, Bury T, Deflandre D, Jerusalem G, Lifrange E, Kaux JF, Crielaard JM, Maquet D. Multidisciplinary rehabilitation program after breast cancer: benefits on physical function, anthropometry and quality of life. Eur J Phys Rehabil Med. 2017 Oct;53(5):633-642. doi: 10.23736/S1973-9087.17.04551-8. Epub 2017 Mar 20. PMID 28322035
- [Background] Demark-Wahnefried W, Rogers LQ, Gibson JT, Harada S, Fruge AD, Oster RA, Grizzle WE, Norian LA, Yang ES, Della Manna D, Jones LW, Azrad M, Krontiras H. Randomized trial of weight loss in primary breast cancer: Impact on body composition, circulating biomarkers and tumor characteristics. Int J Cancer. 2020 May 15;146(10):2784-2796. doi: 10.1002/ijc.32637. Epub 2019 Sep 5. PMID 31442303
- See also: Figures of cancer incidence, prevalence, mortality, survival and risk factors in Spain — http://seom.org/seomcms/images/stories/recursos/Cifras_del_cancer_2020.pdf